CLINICAL TRIAL: NCT06145139
Title: KIDNEY-PAGER: Analysis of Circulating Tumor DNA as a Biomarker in Renal Cancer
Brief Title: KIDNEY-PAGER: Analysis of Circulating Tumor DNA as a Biomarker in Renal Cancer - an Observational Trial
Acronym: KIDNEY-PAGER
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 1-16-02-476-22
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Renal Cancer
Keywords: circulating tumor dna
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall aim of this observational study is to confirm that circulating tumor DNA (ctDNA) detected in plasma and or urine after intended curative treatment for renal cell carcinoma (RCC) can be applied in clinical practice as a marker of subclinical residual disease and risk of recurrence.

DETAILED DESCRIPTION:
OBJECTIVES

The overall objective of the study is to confirm that circulating tumor DNA (ctDNA) detected in plasma and or urine after intended curative treatment for RCC can be applied in clinical practice as a marker of subclinical residual disease and risk of recurrence.

1.1 Primary objectives

1. To confirm that patients with high risk of recurrence can be identified with ctDNA profiling performed immediately after nephrectomy.

   Specifically, we aim to determine in patients with localized RCC (stages I-III) if the three-year disease-free survival is associated with detection of ctDNA in plasma immediately after surgery.

   1.2 Secondary objectives
2. To show that detection of ctDNA pre- and post-operatively can be applied as a risk stratification tool.
3. To validate the potential of a ctDNA-guided follow-up program as compared to the current CT-scan follow-up program. More specifically, to investigate the correlation between ctDNA and CT-scanning findings. The potential is that ctDNA analysis predicts the CT-scan result and can be used to guide when to perform a CT-scan. Potentially, it also adds evidence for the results of CT-scans performed subsequently to an uncertain CT-scan result.
4. To investigate if time to Molecular recurrence using serial ctDNA analysis of longitudinally collected blood samples is shorter than time to Clinical recurrence using standard-of-care radiological imaging surveillance.
5. To find and validate predictive blood- and or tissue-based biomarkers for immunotherapy and or targeted therapies with the aim to identify patients that are more likely to respond to the given therapy administered.
6. To confirm that changes in ctDNA levels reflect the therapeutic effect of the given therapy, such as immunotherapy and or targeted therapies.
7. To delineate markers of tumor aggressiveness and compare to ctDNA measurements

2 INVESTIGATIONAL PLAN

2.1 Overall study design

This study is based on a comprehensive series of blood sampling prospectively and ctDNA analysis performed in RCC patients before and after surgery, during and after treatment, and during surveillance. Patients are followed 5 years from date of surgery.

* Urine, blood sampling and ctDNA analysis pre-operative and immediately after surgery (a postoperative blood sample is drawn on day 14)
* Sampling of tissue from the biopsy and resected specimen as well as adjacent normal.
* Longitudinal blood and urine sampling over a 5-year surveillance period - a blood and urine sample will be drawn simultaneously with the standard-of-care CT-scan-based surveillance program, and from metastatic tissue if a relapse occurs.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a locoregional cancer in the kidney, and with a tumour available for surgical excision, and sufficient performance status for surgery.
* Patients with M1 disease, but no evidence of disease after surgery and local treatment of the metastases.
* Core needle biopsy-proven renal cell carcinoma - all histologic subtypes acceptable, clinical tumour stage I-IV
* Patients 18 years or older
* Patients able to understand and sign written informed consent
* Scheduled for curative intent resectional surgery (partial or radical nephrectomy)

Exclusion Criteria:

* Patients with local disease who are not being offered a nephrectomy.
* Patients who are unlikely to comply with the protocol (e.g. uncooperative attitude), inability to return for subsequent visits and/or otherwise considered by the Investigator to be unlikely to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with curative intent for kidney cancer at Aarhus University Hospital, Denmark.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2033-06-01 (Estimated)

PRIMARY OUTCOMES:
ctDNA can identify high risk patients | baseline, 1 year, 2 year and 3 year
  ctDNA will be determined and levels will be measured, and correlated to relapse status, progression free survival, treatment response and overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Urology Department Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No